CLINICAL TRIAL: NCT04763902
Title: Feasibility and Acceptability of Time Restricted Eating (TRE) Among Native Hawaiian/Pacific Islander Women at Risk for Endometrial Cancer
Brief Title: Time Restricted Eating (TRE) Among Native Hawaiian/Pacific Islander Women at Risk for Endometrial Cancer
Acronym: TIMESPAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Mary Playdon, Assistant Professor, Investigator, University of Utah
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00127142; UL1TR002538 (NIH)
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Trehalase; Appointments and Schedules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating (TRE) Schedule (Experimental): For 8 weeks out of the 14-week randomized dietary crossover study, women will receive prepared frozen lunch and dinner meals as per the control schedule, but will be asked to consume daily meals, snacks, and calories-containing beverages within an 8 to 10-hour period that fits their schedule. The fasting period will ramp up during the first week (Days 1-3, 12-14 h per day, Days 4-6, 14-16 h per day, Days 7+, 16 h per day).
  Interventions: Behavioral: Time Restricted Eating (TRE) Schedule
- Control Schedule (No Intervention): For 4 weeks out of the 14-week randomized dietary crossover study, women will receive prepared frozen lunch and dinner meals, and a standardized breakfast and snacks menu. All meals and snacks will be culturally competent, and meal plans will be individualized to meet weight maintenance energy requirements.

INTERVENTIONS:
Behavioral: Time Restricted Eating (TRE) Schedule — [See arm/group descriptions]
  Arms: Time Restricted Eating (TRE) Schedule

SUMMARY:
The long-term goal of this study is to determine the efficacy of time restricted eating (TRE) for improving metabolic health and preventing endometrial cancer. The primary objective of the protocol is to conduct a 14-week two-arm randomized crossover trial of a dietary intervention to evaluate the feasibility, fidelity and preliminary acceptability of a TRE intervention among Native Hawaiian/Pacific Islander women at risk for developing endometrial cancer, and to provide proof of principle that TRE can improve metabolic health in this population.

DETAILED DESCRIPTION:
Enrollment: The study includes two phases. Phase 1 includes focus groups among 30 Native Hawaiian/Pacific Islander women at risk of endometrial cancer. Focus groups will determine sociocultural influences on (i) dietary behavior including meal timing; (ii) dietary preferences; (iii) proposed meal plans and intervention design; (iv) perceptions of weight loss and body image. In the second study phase, the study team will recruit 10 Pacific Islander women to participate in a 14-week randomized dietary crossover study. Each woman will participate in both intervention arms and act as her own control.

Focus Group: To accomplish all aspects of Aim 1 of this study, the study team will recruit 30 Pacific Islander women at risk for endometrial cancer to conduct virtual focus groups. These focus groups will take place via private videoconference, like Zoom, and a language translator will be provided, as necessary. The focus groups will be attended by a Native Hawaiian/Pacific Islander Community Expert. Questions will be designed to understand sociocultural influences on dietary behavior (questions on social eating, meal timing, and dietary preferences, soliciting feedback on study intervention delivery design, and perceptions of weight loss and body image). An icebreaker will be conducted prior to formal questioning. Sessions will be audio-recorded on the videoconference and an additional device, transcribed verbatim, and checked for accuracy. Two additional team members will be present as note takers. Our Community Expert will be present to help facilitate the session. Questions will be provided at the beginning of the session to ensure cultural sensitivity.

Dietary Intervention: The dietary intervention includes 5 study visits, and features a baseline visit, 2-week run-in period, 4-week control diet schedule, 4-week washout period, and a 4-week, 8 to 10-hour Time Restricted Eating (TRE) protocol (8 to 10-hour feeding and 14 to 16-hour fasting periods). A follow-up questionnaire will be mailed 6-months post- intervention. For the control schedule, women will receive frozen lunch and dinner meals and a standardized breakfast and snacks menu. All meals and the breakfast/snack menu will be designed to be culturally competent with feedback from the focus groups, and meal plans will be individualized to meet weight maintenance energy requirements. For the TRE schedule, women will receive prepared frozen lunch and dinner meals as per the control schedule, but will be asked to consume daily meals, snacks, and calorie-containing beverages within an 8 to 10-hour period that fits their schedule. They will be asked to maintain their regular sleep and physical activity schedule. The fasting period will ramp up during the first week (Days 1-3, 12-14 h per day, Days 4-6, 14-16 h per day, Days 7+, 16 h per day). Women will be asked to schedule the eating period at the same time each day. All meals (control and TRE) will be provided by the Metabolic Kitchen located at the University of Utah.

Visit 1: During the baseline visit, a coordinator will obtain consent from the participant, and they will be asked to compete questionnaires asking about clinical and demographic factors, chronotype, and physical activity, and various anthropometric measurements will be taken. Following the baseline visit, participants will undergo a 2-week run-in period. During this time, the goal is to record women's usual times of eating episodes and appetite while following their habitual diet.

Visit 2: Women will provide fasting blood and stool samples, and anthropometric measurements will be taken. Following visit 2, participants will undergo the control or TRE schedule for 4 weeks.

Visit 3: After 4 weeks, participants will undergo visit 3 and will be asked to provide fasting blood and stool samples, and anthropometric measures will be taken. Following visit 3, participants will undergo a 4-week washout period, where women are able to return to their usual lifestyle.

Visit 4: Visit 4 will occur after the 4-week washout period, and will include a telephone consultation to discuss the next study phase and schedule meal provision. For the following 4-weeks, participants will then undergo the opposite feeding schedule (either control or TRE).

Visit 5: During the final visit, women will provide fasting blood and stool samples, and anthropometric measures will be taken.

During the run-in period, the TRE phase and the control phase, participants will record timing of eating episodes using the MyCircadian Clock phone app, complete 3 x 24-hour diet recalls, a single physical activity recall, and 7-days of sleep and physical activity will be objectively measured using an Actiwatch device. Hunger and satiety will be evaluated at random through the MyCircadian Clock phone app.

A study exit interview will be conducted via Zoom conference call to debrief on the intervention and obtain detailed information on acceptability of the protocol. Approximately 6-months after the end of the intervention period, women will complete a mailed follow-up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

All Aims:

* Native Hawaiian/Pacific Islander females aged 18 years or older
* Overweight or obese (BMI>25kg/m2) OR have a history of non-insulin dependent diabetes OR have a history of complex atypical endometrial hyperplasia
* Have a working cell phone that can download an App
* Able to use cell phone during day (e.g. at work)
* Not a night shift worker

Applicable Only to Aims 2 & 3:

* Able to attend study visits at the Huntsman Cancer Institute Center for HOPE

Exclusion Criteria:

All Aims:

* Unable to provide informed consent

Applicable Only to Aims 2 & 3:

* Necessity of a special diet that precludes adjustment of meal timing and/or macronutrient content
* Have a history of insulin dependent diabetes
* Have a history of hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Women Referred that are Consented | From baseline to Visit 5 (Week 14)
  Feasibility of the TRE intervention will be measured by calculating a proportion (%) of women who were referred that were consented into the study. The study will be considered feasible if > 70% of participants are consented and retained.
Attrition as a Function of Time | From baseline to Visit 5 (Week 14)
  Number of participants who withdraw throughout the course of the study.
Percent of Scheduled Assessments Completed | From baseline to Visit 5 (Week 14)
  Feasibility of the TRE intervention will be assessed by calculating a percentage of scheduled biospecimen collection and questionnaires completed.
Number of TRE-Adherent Days per Week | From baseline to Visit 5 (Week 14)
  Feasibility of the TRE intervention will be measured by calculating the number of TRE-adherent days per week. Participants will be considered adherent if they fasted between 14-18 hours per day during the TRE phase according to a mealtime log. The study will be considered feasible if women adhere to the TRE protocol on average 5 days per week.
Percentage of Meals Delivered On Schedule | From baseline to Visit 5 (Week 14)
  Feasibility of the TRE intervention will be measured by calculating a percentage of meals delivered on schedule.
Fidelity of Time Restricted Eating (TRE) Intervention | From baseline to Visit 5 (Week 14)
  Fidelity will be evaluated as a percentage of protocol checklist items delivered as intended with a goal of 90%.

SECONDARY OUTCOMES:
Change in blood pressure assessed via electronic blood pressure monitor | Baseline (Visit 1), Visit 2 (Week 2), Visit 3 (Week 6), Visit 5 (Week 14)
  Blood pressure will be taken using an electronic blood pressure monitor.
Change in waist circumference assessed via measuring tape | Baseline (Visit 1), Visit 2 (Week 2), Visit 3 (Week 6), Visit 5 (Week 14)
  Waist circumference will be measured using a measuring tape.
Change in BMI assessed via height and weight | Baseline (Visit 1), Visit 2 (Week 2), Visit 3 (Week 6), Visit 5 (Week 14)
  Participants' height and weight will be taken and used to calculate BMI.
Change in fasting blood glucose assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6), Visit 5 (Week 14)
  A small sample of blood will be taken from participants at designated study visits.
Change in HOMA-IR assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6), Visit 5 (Week 14)
  A small sample of blood will be taken from participants at designated study visits.
Change in c-peptide assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6), Visit 5 (Week 14)
  A small sample of blood will be taken from participants at designated study visits.
Change in triglycerides assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6), Visit 5 (Week 14)
  A small sample of blood will be taken from participants at designated study visits.
Change in HDL-cholesterol assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6), Visit 5 (Week 14)
  A small sample of blood will be taken from participants at designated study visits.
Change in high sensitivity C-reactive protein assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6), Visit 5 (Week 14)
  A small sample of blood will be taken from participants at designated study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Playdon, PhD, MPH, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No